CLINICAL TRIAL: NCT01290068
Title: Visual Outcomes After Bilateral Surgical Cataract Phacoemulsification: AcrySof® ReSTOR IOL Implantation Compared to Monofocal IOL Implantation
Brief Title: Visual Outcomes After Cataract Surgery: Multifocal AcrySof® IQ ReSTOR® Intraocular Lenses Versus Monofocal Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDG-10-269
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-03

CONDITIONS: Cataract
Keywords: Intraocular Lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- ReSTOR +3 (Experimental): AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL, bilateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL
- ReSTOR +3 Toric (Experimental): AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative corneal astigmatism, bilateral implantation, or implanted in 1 eye with AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL in the other eye
  Interventions: Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL; Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL
- Monofocal (Active Comparator): Monofocal IOL, bilateral implantation
  Interventions: Device: Monofocal IOL

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL — Multifocal IOL with extended secondary focal point implanted for long-term use over the lifetime of the cataract patient
  Other Names: SN6AD1
  Arms: ReSTOR +3; ReSTOR +3 Toric
Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL — Multifocal IOL with extended secondary focal point and astigmatism correction implanted for long-term use over the lifetime of the cataract patient
  Other Names: SND1T2, SND1T3, SND1T4, SND1T5
  Arms: ReSTOR +3 Toric
Device: Monofocal IOL — Monofocal IOL implanted for long-term use over the lifetime of the cataract patient
  Arms: Monofocal

SUMMARY:
The purpose of this study is to assess and compare visual outcomes of the AcrySof® IQ ReSTOR® +3.0 D intraocular lens (IOL) to a commercially available monofocal IOL in cataract patients.

DETAILED DESCRIPTION:
This study included subjects with bilateral age-related cataracts and either no preoperative corneal astigmatism, or preoperative regular corneal astigmatism confirmed by autokeratometry of ≤2.5 D.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign an Informed Consent;
* Willing and able to attend post-operative examinations as per protocol schedule;
* Diagnosis of bilateral, age-related cataracts;
* Planned cataract removal via phacoemulsification with implantation of an IOL;
* Available to undergo second eye surgery within 6 weeks of the first eye surgery;
* Fulfill the recommendations of the "Warnings" and "Precautions" sections of the AcrySof IQ ReSTOR IOL and Monofocal IOL package inserts;
* No preoperative corneal astigmatism or preoperative regular corneal astigmatism ≤2.5D;
* Qualify in both eyes for either AcrySof® IQ ReSTOR® IOL Model SN6AD1 or AcrySof® IQ ReSTOR® Toric IOL Models SND1T2 through SND1T5 as indicated by the AcrySof IQ ReSTOR Multifocal Toric web-based calculator;
* Able to read and understand one of the following languages: Dutch, French, German, Italian, Spanish, English or Catalan.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Previous corneal surgery and/or reshaping;
* Any abnormality, disease and/or conditions of the cornea (ie, keratoconus, corneal dystrophy, severe keratitis, corneal scar, etc.), which would clinically contraindicate the implantation of a toric IOL;
* Planned multiple procedures during cataract/IOL implantation surgery;
* Planned limbal relaxing incisions, excimer laser treatment or similar procedures prior to or during the course of the study;
* Pregnant, lactating, or planning pregnancy during the course of study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brand Lead, Surgical, Global Medical Affairs, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 20 investigative sites located in France (3), Germany (4), Great Britain (1), Italy (3), Netherlands (4), and Spain (5).
Pre-assignment Details: This reporting group includes all randomized participants, as randomized.
Groups:
- Multifocal IOL: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL, with or without astigmatism correction, bilateral implantation
- Monofocal IOL: Monofocal IOL, bilateral implantation
Period: Overall Study
Arm/Group | Multifocal IOL | Monofocal IOL
Started | 108 | 100
Implanted | 108 | 98
Completed | 101 | 94
Not Completed | 7 | 6
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by subject prior to implant | 0 | 2
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants to whom the randomized IOL was presented and/or implanted during the first eye surgery (from a try to a full success), as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Multifocal IOL | Monofocal IOL | Total
Number analyzed (Participants) | 108 | 98 | 206
Age, Customized [Number; unit: participants]
  21 to 59 years | 13 | 7 | 20
  60 to 69 years | 40 | 36 | 76
  70 to 79 years | 40 | 45 | 85
  ≥80 years | 15 | 10 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 58 | 121
  Male | 45 | 40 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Classified as Responders
Description: Distance VA and near VA were measured binocularly (both eyes together) without visual correction using ETDRS (Early Treatment of Diabetic Retinopathy Study) charts positioned at a consistent, manufactured distance. VA was measured in logMAR (logarithm of the minimum angle of resolution), with a lower logMAR value indicating better visual acuity. A responder was defined as a participant who achieved bilateral uncorrected distance visual acuity and bilateral uncorrected near visual acuity of ≤0.1 LogMAR at the Month 6 visit.
Time Frame: Month 6 after second eye implantation
Population: This analysis population includes all randomized participants to whom the randomized IOL was presented and/or implanted during the first eye surgery (from a try to a full success), as randomized. Last observation carried forward (LOCF) was used for missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 105 | 97
percentage of participants | 45.7 | 2.1

2. Primary Outcome: Proportion of Participants Reporting Spectacle Independence at All Distances
Description: Spectacle independence at all distances; ie, where type of spectacles used/prescribed equaled 'No spectacles', was evaluated. If for the 6-month visit, spectacle type information was missing for the spectacle independence endpoint, but the subject attended this 6-month visit, subject was assumed to be spectacle independent.
Time Frame: Month 6 after second eye implantation
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 101 | 95
percentage of participants | 73.3 | 25.3

3. Primary Outcome: Mean Vision-Related Quality of Life as Reported on the NEI-RQL 42 (5 Dimensions)
Description: Vision-related quality of life dimensions were evaluated using the National Eye Institute Refractive Error Quality of Life instrument (NEI-RQL 42), a self-administered questionnaire. Each dimension was scored between 0 to 100, with a higher score indicating a better vision-related Quality of Life. 5 of the dimensions were prespecified as primary.
Time Frame: Month 6 after second eye implantation
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 108 | 98
units on a scale
  Near vision: number analyzed (Participants) | 100 | 93
  Near vision | 87.63 (1.868) | 83.57 (1.951)
  Activity limitations: number analyzed (Participants) | 99 | 90
  Activity limitations | 95.19 (1.431) | 94.85 (1.511)
  Dependence on correction: number analyzed (Participants) | 99 | 92
  Dependence on correction | 83.67 (3.512) | 46.34 (3.686)
  Appearance: number analyzed (Participants) | 98 | 90
  Appearance | 84.48 (2.723) | 76.79 (2.875)
  Satisfaction with correction: number analyzed (Participants) | 98 | 90
  Satisfaction with correction | 84.81 (2.071) | 82.40 (2.179)

4. Secondary Outcome: Median Total Spectacle Cost Prior to Any Reimbursement
Description: Total spectacle cost includes the frame, lens, and any reimbursement from national health systems or private insurance. Costs collected in pounds sterling were converted to euros.
Time Frame: Month 6 after second eye implantation
Population: This analysis population includes all randomized and implanted participants. If total cost was missing for a spectacle independent subject, €0 was imputed. If total cost was missing for a spectacle-dependent subject, mean cost for all spectacle dependent-subjects in that group with a known total cost for the same type of spectacles was imputed.
Measure: Median (Inter-Quartile Range); unit: euros
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 101 | 95
euros | 0.00 [0.00 to 8.50] | 85.729 [0.00 to 147.42]

ADVERSE EVENTS:
Time Frame: An Adverse Event (AE) was defined as any untoward medical occurrence in a subject, user, or other persons regardless of causal relationship to the device.
Description: This reporting group includes all randomized subjects with at least 1 implanted IOL, as implanted. Note: 3 subjects randomized to Multifocal received Monofocal instead, and 1 subject randomized to Monofocal received Multifocal.
Arm/Group | Multifocal IOL | Monofocal IOL
Serious Adverse Events (participants affected / at risk) | 13/106 | 9/100
Other Adverse Events (participants affected / at risk) | 0/106 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multifocal IOL (N=106) | Monofocal IOL (N=100)
Cardiac disorder (Cardiac disorders) | 1 | 0
Astigmatism (Eye disorders) | 1 | 0
Corneal oedema (Eye disorders) | 1 | 0
Cystoid macular oedema (Eye disorders) | 1 | 0
Iridocele (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Posterior capsular opacification (Eye disorders) | 2 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 1
Vitreous loss (Eye disorders) | 1 | 0
Vitritis (Eye disorders) | 0 | 1
Intestinal functional disorder (Gastrointestinal disorders) | 1 | 0
Device material issue (General disorders) | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0
Eye operation complication (Injury, poisoning and procedural complications) | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Chronic pulmonary obstructive disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.